CLINICAL TRIAL: NCT04074733
Title: Diagnostic Performance of the Ultra Low-Dose (ULD) Scanner vs. Diagnostic Performance With Standard X-rays in the Emergency Department Compared With Performance of the Standard Classical-dose Scanner for Trauma of the Dorsolumbar Spine, Pelvis and Extremities
Acronym: ULD-Traumato
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRCi/2018/AL-01; 2019-A00472-55 (Other: ANSM)
Record Dates: First submitted 2019-08-23; First posted 2019-08-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Bone Fractures
Keywords: ULD
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with fractures
  Interventions: Diagnostic Test: Patient undergoes a ULD scan; Diagnostic Test: Patient undergoes a standard X-ray; Diagnostic Test: Patient undergoes a classic-dose scan

INTERVENTIONS:
Diagnostic Test: Patient undergoes a ULD scan — The following doses will be applied:
  6 mGy.cm for the extremities 50 mGy.cm for the dorsal spine 130 mGy.cm for the lumbar spine 130 mGy.cm for the pelvis
Diagnostic Test: Patient undergoes a standard X-ray — The following doses will be applied:
  For the pelvis : front view and profile for the hip. For the dorsal spine : front and profile. For the lumbar spine : front and profile For the extremities : front and profile
Diagnostic Test: Patient undergoes a classic-dose scan — The following doses will be applied:
  6 mGy.cm for the extremities 50 mGy.cm for the dorsal spine 130 mGy.cm for the lumbar spine 130 mGy.cm for the pelvis

SUMMARY:
The conventional standard-dose scanner leads to a significantly greater X-ray exposure than the standard X-ray. Recently, technological innovations like the ULD ("Ultra Low Dose") scanner have been developed to reduce the dose of X-rays delivered to the patient. The general purpose of this study is to validate the ULD scanner in case of emergency trauma of the dorsolumbar spine, pelvis and / or extremities.

DETAILED DESCRIPTION:
The main purpose of this study is to compare the diagnostic performances of the ULD scanner with those of the standard X-ray when looking for fractures of the dorsolumbar region, the pelvis, proximal femur or the extremities, in an emergency situation in adults, once the diagnosis of fracture has been ascertained by the classical standard-dose scanner (gold standard). The statistical analyses will be performed with the help version 9.4 or subsequent versions of SAS software (SAS Institute, Cary, NC, USA) and/or version 3.5.1 or subsequent versions of R software (R Development Core Team (2018). R Foundation for Statistical Computing, Vienna, Austria).

The secondary objectives of this study are to:

A. Compare the diagnostic performances of the two examination methods under study (ULD scan vs. standard X-ray) in the search for bone structure anomalies, damage to the soft tissues, damage to the joints and/or discopathies at the site(s) involved.

B. Compare the diagnostic performances of the two examination methods under study) (ULD scan vs. standard X-ray) in the search for fractures of the site involved. C. Evaluate the diagnostic agreement between two readers (senior radiologist and junior radiologist) for each of the two examination methods under study (ULD scan vs. standard X-ray).

D. Compare the radiologist's self-declared impression of each of the two examination methods under study (ULD scan vs. standard X-ray) in terms of subjective quality: overall image quality, diagnostic quality of the examination method and the level of confidence in the diagnosis made, overall and for each of the two readers (senior and junior).

E. Compare the doses of X-rays administered for each of the two examination methods under study (ULD scan vs. standard X-ray).

F. Compare the interpretation time for each examination method under study (ULD scan vs. standard X-ray), globally and for each of the two readers (senior and junior).

For the evaluation of the diagnostic performances (main objective and secondary objectives A et B), only the senior radiologist's interpretation will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a BMI <40 kg / m²
* Emergency department patient for trauma of the dorso-lumbar spine, pelvis, proximal femurs, and / or extremities requiring standard radiographs
* Patient with painful symptomatology causing suspicion of a broken bone
* Patient or family member / trusted person / family member who has given free and informed consent
* Patient or family member / trusted person / family member who has signed the consent form
* Patient beneficiary or affiliate of a health insurance plan

Exclusion criteria:

* Patient participating in a category 1 study
* Patient in a period of exclusion determined by another study
* Patient on under juridical protection, under curatorship or under guardianship
* Patient for whom it is impossible to give informed information
* Pregnant, parturient or nursing patient
* Polytraumatised patient
* Patients in vital emergency requiring urgent scanner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient presenting at the emergency department patient for trauma of the dorso-lumbar spine, pelvis, proximal femurs, and / or extremities requiring standard X-rays.
Sampling Method: Non-Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Presence of at least one fracture in the dorsal spine evaluated with a classical, standard-dose scan (Gold standard) | Day 0
  YES/NO
Presence of at least one fracture in the lumbar spine evaluated with a classical, standard-dose scan (Gold standard) | Day 0
  YES/NO
Presence of at least one fracture of the pelvis and proximal femurs evaluated with a classical, standard-dose scan (Gold standard) | Day 0
  YES/NO
Presence of at least one fracture of the hands / wrists evaluated with a classical, standard-dose scan (Gold standard) | Day 0
  YES/NO
Presence of at least one fracture of the feet /ankles evaluated with a classical, standard-dose scan (Gold standard) | Day 0
  YES/NO
Presence of at least one fracture in the dorsal spine evaluated with a ULD scan | Day 0
  YES/NO
Presence of at least one fracture in the lumbar spine evaluated with a ULD scan | Day 0
  YES/NO
Presence of at least one fracture in the pelvis and proximal femurs evaluated with a ULD scan | Day 0
  YES/NO
Presence of at least one fracture of the hands / wrists evaluated with a ULD scan | Day 0
  YES/NO
Presence of at least one fracture of the feet /ankles evaluated with a ULD scan | Day 0
  YES/NO
Presence of at least one fracture of the dorsal spine evaluated with a standard X-ray | Day 0
  YES/NO
Presence of at least one fracture of the lumbar spine evaluated with a standard X-ray | Day 0
  YES/NO
Presence of at least one fracture of the pelvis and proximal femurs evaluated with a standard X-ray | Day 0
  YES/NO
Presence of at least one fracture of the hands / wrists evaluated with a standard X-ray | Day 0
  YES/NO
Presence of at least one fracture of the feet /ankles evaluated with a standard X-ray | Day 0
  YES/NO

SECONDARY OUTCOMES:
Presence of an abnormality of the bone structure at the anatomic site(s) concerned evaluated with a classical Gold Standard scan | Day 0
  YES/NO
Presence of an abnormality of the soft tissues at the anatomic site(s) concerned evaluated with a classical Gold Standard scan | Day 0
  YES/NO
Presence of an abnormality of the joints at the anatomic site(s) concerned evaluated with a classical Gold Standard scan | Day 0
  YES/NO
Presence of an abnormality of the invertebral discs at the anatomic site(s) concerned evaluated with a classical Gold Standard scan | Day 0
  YES/NO
Presence of an abnormality of the bone structure at the anatomic site(s) concerned evaluated with a ULD scan | Day 0
  YES/NO
Presence of an abnormality of the soft tissues at the anatomic site(s) concerned evaluated with a ULD scan | Day 0
  YES/NO
Presence of an abnormality of the joints at the anatomic site(s) concerned evaluated with a ULD scan | Day 0
  YES/NO
Presence of an abnormality of the invertebral discs at the anatomic site(s) concerned evaluated with a ULD scan | Day 0
  YES/NO
Presence of an abnormality of the bone structure at the anatomic site(s) concerned evaluated with a standard X-ray | Day 0
  YES/NO
Presence of an abnormality of the soft tissues at the anatomic site(s) concerned evaluated with a standard X-ray | Day 0
  YES/NO
Presence of an abnormality of the joints at the anatomic site(s) concerned evaluated with a standard X-ray | Day 0
  YES/NO
Presence of an abnormality of the intervertebral discs at the anatomic concerned site(s) evaluated with a standard X-ray | Day 0
  YES/NO
Image quality of the ULD scanner and standard X-ray | Day 0
  By means of a 4-point Likert scale, both the senior and junior radiologists can give their subjective impression of the overall image quality of each of the two examination methods under study (ULD scan vs. standard X-ray) by saying how much they agree or disagree that the overall quality of the image is good enough to detect a fracture. On the Lickert scale, 1- Uninterpretable, 2- Interpretable in spite of a slight technical problem (centering, movement, constant), 3-Completely interpretable in spite of a slight technical problem. 4- No technical problem.
Diagnostic quality of the ULD scanner and standard X-ray | Day 0
  Using a 5-point Lickert scale (in which 1= Inacceptable, 2 = Sub-optimal, 3 = Acceptable, 4 = Above average, 5- Excellent) both the senior and junior radiologists will give their subjective impression of the overall diagnostic quality of each of the two examination methods under study (ULD scan vs. standard X-ray).
Confidence level of the ULD scanner and standard X-ray | Day 0
  Using a 5-point Lickert scale (1- Very poor, 2- Poor, 3- Fair, 4- Good, 5- Excellent) both the senior and junior radiologists will give their subjective impression of their overall level of confidence in the diagnosis made for each of the two examination methods under study (ULD scan vs. standard X-ray).
Effective dose for each exam with the ULD scanner | Day 0
  No. of millisieverts (mSv)
Effective dose for each exam with the standard X-ray | Day 0
  No. of millisieverts (mSv)
Interpretation time for each exam with the ULD scanner | Day 0
  Measured in minutes
Interpretation time for each exam with the standard X-ray | Day 0
  Measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed LARBI, Dr., Principal Investigator — CHU de Nîmes (Nîmes University Hospital)
Locations (5):
- France (5):
  - Centre Hospitalier Universitaire, Nîmes, Gard
  - Clinique de l'Union, Saint-Jean, Haute-Garonne
  - Clinique du Parc, Castelnau-le-Lez, Hérault
  - Centre Hospitalier de Mont-de-Marsan, Mont-de-Marsan, Nouvelle-Aquitaine
  - Menouer TALEB, Alès

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hamard A, Greffier J, Bastide S, Larbi A, Addala T, Sadate A, Beregi JP, Frandon J. Ultra-low-dose CT versus radiographs for minor spine and pelvis trauma: a Bayesian analysis of accuracy. Eur Radiol. 2021 Apr;31(4):2621-2633. doi: 10.1007/s00330-020-07304-8. Epub 2020 Oct 9. PMID 33034747